CLINICAL TRIAL: NCT02367482
Title: Tryptophan Metabolism in Human Brain Tumors: For Patients Whose Clinical Treatment Includes NovoTTF
Brief Title: Tryptophan Metabolism in Human Brain Tumors-Novocure
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Csaba Juhasz, Principal Investigator, Wayne State University
Other Study IDs: Novocure rGBM AMT-PET
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma
Keywords: rGBM; Recurrent GBM; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — we will collect and analyze the tumor specimens obtained prior to NovoTTF therapy (as well as any tissue specimens available if a patient undergoes surgical resection after initiating NovoTTF therapy) for various histopathologic features (e.g., proliferative activity, vessel density, expression of L-type amino acid transporter), and correlate with neuroimaging findings and clinical response to NovoTTF. This may provide additional useful information on potential mechanisms of treatment failure.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NovoTTF: NovoTTF treatment will be administered as usual during the imaging study either in monotherapy or in combination with other treatments (initiated prior to NovoTTF therapy). The treatment plan or intervention will not be altered in any way. Two AMT-PET scans will be added to the management scheme: a baseline PET shortly before and a follow-up PET scan 2-3 months after the start of NovoTTF treatment.

SUMMARY:
In this research study, we will track the build-up of tryptophan, a radioactive tracer, in the brain using positron emission tomography (PET) scanning. Tryptophan, in its natural state, is an amino acid (one of the building blocks of proteins) that is normally present in the brain, and is used by the brain cells to create various other compounds. This process is altered in the presence of a brain tumor. By using a form of tryptophan marked with a small amount of radiation, we will be able to track this process during the course of the PET scan. This research will help determine if AMT PET is a useful method to recognize and differentiate between various types of brain tumors. In addition, to study the mechanisms of altered tryptophan uptake in the tumor and brain, we will also measure tryptophan levels and related molecules in your blood (obtained as a part of the PET procedure) and tumor tissue (in case you will have surgery to remove the tumor). This will help us to find new approaches to treat brain tumors in the future by altering abnormal tryptophan metabolism.

DETAILED DESCRIPTION:
If you agree to take part in this research study, you will be asked to have:

1. A PET scan, 2. brief clinical questionnaires, and 3. biochemical studies of blood and tumor tissue. You will also have a second PET scan later, 2-3 months after the start of NovoTTF therapy, to determine if there are changes in the tumor that can be detected by PET. Your ability to participate in the study will be based, in part, on the results of the magnetic resonance images (MRI) in your medical chart from earlier clinical procedures. Once we receive the results of the PET scan, these will be compared to the MRI in order to help us analyze the tryptophan uptake in your brain. It will take about 3 hours to complete the PET scan; this includes the completion of the questionnaire, preparation and scanning. The actual scanning time will be 70 minutes. If you are a female of child-bearing age, we will need a small urine sample from you before starting the PET scanning procedure to make absolutely sure that you do not have unknown pregnancy for which radiation exposure might be harmful.

1. The PET scan will be used to measure the accumulation of the injected radioactive tracer AMT in your brain. To make this measurement more accurate, we will use your clinically obtained MRI scan(s), which was used to diagnose the tumor, to identify the exact location and extent of the tumor. For the PET scan, an intravenous catheter (a small tube placed in your vein) will be inserted for the injection of the AMT for this PET scan. It is the tracer that the PET scanner "sees" when performing the scan. The amount of the tracer, which will be given is very small (5 ml, the volume of a teaspoon), and therefore no side effects are expected from the tracer itself. A second intravenous catheter will be inserted to collect blood samples during the scan; a total of less than 2 teaspoons of blood will be collected. Participants may be sedated (put into sleep with some medicine) if they are unable to remain still for the scanning period.
2. On the day of the PET scan, we will ask you to fill out a brief clinical questionnaire, and also an additional multiple-choice questionnaire to screen for potential mood problems (which often coincide with brain tumors). Participants with a potential speech (comprehension) problem will also be administered a brief speech test. The goal of these tests is to identify various clinical problems that can be associated with brain tumors and affected by abnormal tryptophan metabolism that we measure with the PET scan.
3. If you have surgery to remove the tumor, a portion of the removed tissue will be used for biochemical studies. The doctor will not remove more tissue than needed for your care. The blood (obtained during the PET scanning) and tumor tissue (obtained during surgery) will be processed for analysis and stored in a locked container or freezer in a laboratory. In addition, we will review the clinical pathology report, so that we can correlate your PET results to type and grade of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and MRI diagnosis of recurrent GBM.
2. Age ≥22 years.
3. Patient agrees to NovoTTF treatment but has not started treatment yet.
4. Patient agrees to undergo a baseline and a follow-up AMT-PET scan during NovoTTF treatment.
5. Patient able to provide informed consent.

Exclusion Criteria:

1. Resective surgery within 2 months prior to the initial AMT-PET scan (acute/subacute post-surgical inflammatory changes may cause false positive increased uptake on AMT-PET).
2. Severe increased intracranial pressure, status epilepticus, or other severe complications of the tumor, requiring emergency or urgent intervention.
3. Positive pregnancy test (because of radiation involved in PET scanning).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible and agreeable to undergo NovoTTF treatment at KCC/WSU due to recurrent glioblastoma (initial or subsequent tumor recurrence) will be recruited by the multidisciplinary neuro-oncology team to undergo the two AMT-PET studies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Interval Changes of Tumoral Metabolism | 2-3 months
  To measure interval changes of tumoral metabolism, blood flow, and metabolites (NAA, choline, creatine, lipid, lactate) using AMT-PET, perfusion MRI, and 1H-MRS, respectively, in patients with recurrent GBM treated with NovoTTF.

SECONDARY OUTCOMES:
Interval changes of tumoral tryptophan metabolism | 2-3 months
  To evaluate if interval changes of tumoral tryptophan metabolism, perfusion, and/or metabolites as well as histopathologic features (e.g., blood vessel density) have a predictive value for progression-free and overall survival in patients treated with NovoTTF.

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Juhasz, MD, PhD, Principal Investigator — Wayne State University; Sandeep Mittal, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No